CLINICAL TRIAL: NCT03410771
Title: Bioelectrical Impedance Analysis as a Bedside Tool to Estimate Volume of Distribution of Hydrophilic Antimicrobials in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Matthias Gijsen, PharmD PhD researcher - Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: mp05488
Record Dates: First submitted 2018-01-08; First posted 2018-01-25 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Electric Impedance; Pharmacokinetics; Capillary Leak Syndrome
Keywords: Distribution Volume; Antibiotics
MeSH Terms: conditions — Capillary Leak Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ICU patients on amoxicillin/clavulanic acid
  Interventions: Drug: Monitor antibiotic exposure (PK profile); Device: Bioelectrical impedance analysis to measure body composition
- ICU patients on piperacillin/tazobactam
  Interventions: Drug: Monitor antibiotic exposure (PK profile); Device: Bioelectrical impedance analysis to measure body composition
- ICU patients on meropenem
  Interventions: Drug: Monitor antibiotic exposure (PK profile); Device: Bioelectrical impedance analysis to measure body composition
- ICU patients on vancomycin
  Interventions: Drug: Monitor antibiotic exposure (PK profile); Device: Bioelectrical impedance analysis to measure body composition

INTERVENTIONS:
Drug: Monitor antibiotic exposure (PK profile) — several plasma samples to measure drug exposure
Device: Bioelectrical impedance analysis to measure body composition — non invasive analysis (electrodes) to measure extra- and intracellular, and total body water.

SUMMARY:
Bioelectrical impedance analysis is studied as a bedside tool to estimate capillary leak in order to guide dosing of hydrophilic antimicrobials.

DETAILED DESCRIPTION:
Abstract Background: Recent data suggest that antimicrobial pharmacokinetics (PK) like volume of distribution (Vd) or drug clearance (CL) is extremely altered in critically ill patients with sepsis or septic shock due to pathophysiological alterations (e.g. influence on fluid status). Bioelectrical impedance analysis (BIA) was recently introduced as a simple, non-invasive, bedside technique to assess hydration status. The primary aim of the present study was to explore the correlation between BIA parameters and Vd of hydrophilic antimicrobial agents in critically ill patients. Furthermore, the relationship between BIA measurements and clinical observations was evaluated.

Methods: We performed a validation study in healthy volunteers in September 2015 that confirmed the reproducibility of BIA. Subsequently, a prospective observational study was carried out in eligible patients treat-ed with amoxicillin/clavulanic acid, meropenem, piperacillin/tazobactam or vancomycin, admitted at the in-tensive care unit (ICU) of the University Hospitals Leuven from October 2015 to March 2016. BIA measurement was performed on the same day as the collection of blood samples to calculate PK parameters of the administered antibiotic.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to ICU ward
* Treated with one of the four studied antimicrobials

Exclusion Criteria:

* <18 years
* Pregnant
* Do Not Resuscitate code 2 or 3
* Renal replacement therapy
* ECMO
* Pacemaker/defibrillator
* Extended burns or dermatological ilness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to our intensive care unit
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Correlation between BIA parameters and Vd of hydrophilic antimicrobial agents | 6-12 hours (= dosing interval) depending on the antimicrobial studied
  Extracellular water (ECW), intracellular water, total body water (TBW), all expressed in liter, and ECW expressed as % of TBW will be correlated with Vd (L/kg) of vancomycin, meropenem, amoxicillin/clavulanic acid and piperacillin/tazobactam

SECONDARY OUTCOMES:
Correlation between BIA assessed hydration status and clinical observations | 1 day
  Hydration status measured by BIA (dehydrated, normohydrated, hyperhydrated) will be correlated with SOFA score and cumulative fluid balance (L)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Spriet, PharmD PhD, Study Director — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
To be determined

REFERENCES:
- [Background] Jones SL, Tanaka A, Eastwood GM, Young H, Peck L, Bellomo R, Martensson J. Bioelectrical impedance vector analysis in critically ill patients: a prospective, clinician-blinded investigation. Crit Care. 2015 Aug 12;19(1):290. doi: 10.1186/s13054-015-1009-3. PMID 26260579
- [Background] Balik M, Sedivy J, Waldauf P, Kolar M, Smejkalova V, Pachl J. Can bioimpedance determine the volume of distribution of antibiotics in sepsis? Anaesth Intensive Care. 2005 Jun;33(3):345-50. doi: 10.1177/0310057X0503300310. PMID 15973917
- [Background] Malbrain ML, Huygh J, Dabrowski W, De Waele JJ, Staelens A, Wauters J. The use of bio-electrical impedance analysis (BIA) to guide fluid management, resuscitation and deresuscitation in critically ill patients: a bench-to-bedside review. Anaesthesiol Intensive Ther. 2014 Nov-Dec;46(5):381-91. doi: 10.5603/AIT.2014.0061. PMID 25432557
- [Background] Dewitte A, Carles P, Joannes-Boyau O, Fleureau C, Roze H, Combe C, Ouattara A. Bioelectrical impedance spectroscopy to estimate fluid balance in critically ill patients. J Clin Monit Comput. 2016 Apr;30(2):227-33. doi: 10.1007/s10877-015-9706-7. Epub 2015 May 29. PMID 26018457
- [Background] Lee YH, Lee JD, Kang DR, Hong J, Lee JM. Bioelectrical impedance analysis values as markers to predict severity in critically ill patients. J Crit Care. 2017 Aug;40:103-107. doi: 10.1016/j.jcrc.2017.03.013. Epub 2017 Mar 22. PMID 28380407
- [Background] Samoni S, Vigo V, Resendiz LI, Villa G, De Rosa S, Nalesso F, Ferrari F, Meola M, Brendolan A, Malacarne P, Forfori F, Bonato R, Donadio C, Ronco C. Impact of hyperhydration on the mortality risk in critically ill patients admitted in intensive care units: comparison between bioelectrical impedance vector analysis and cumulative fluid balance recording. Crit Care. 2016 Apr 8;20:95. doi: 10.1186/s13054-016-1269-6. PMID 27060079
- [Background] Roberts JA, Abdul-Aziz MH, Lipman J, Mouton JW, Vinks AA, Felton TW, Hope WW, Farkas A, Neely MN, Schentag JJ, Drusano G, Frey OR, Theuretzbacher U, Kuti JL; International Society of Anti-Infective Pharmacology and the Pharmacokinetics and Pharmacodynamics Study Group of the European Society of Clinical Microbiology and Infectious Diseases. Individualised antibiotic dosing for patients who are critically ill: challenges and potential solutions. Lancet Infect Dis. 2014 Jun;14(6):498-509. doi: 10.1016/S1473-3099(14)70036-2. Epub 2014 Apr 24. PMID 24768475
- [Background] Basso F, Berdin G, Virzi GM, Mason G, Piccinni P, Day S, Cruz DN, Wjewodzka M, Giuliani A, Brendolan A, Ronco C. Fluid management in the intensive care unit: bioelectrical impedance vector analysis as a tool to assess hydration status and optimal fluid balance in critically ill patients. Blood Purif. 2013;36(3-4):192-9. doi: 10.1159/000356366. Epub 2013 Dec 20. PMID 24496190